CLINICAL TRIAL: NCT00247208
Title: The SOS (Stenting Of Saphenous Vein Grafts) Randomized-controlled Trial of a Paclitaxel-eluting Stent vs. a Bare Metal Stent in Saphenous Vein Graft Lesions
Brief Title: The SOS (Stenting Of Saphenous Vein Grafts) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Clark R. Gregg Fund, Harris Methodist Foundation (Unknown); University of Arkansas (Other); US Department of Veterans Affairs (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Southern Arizona VA Health Care System (U.S. Federal Agency); Onassis Cardiac Surgery Centre (Other)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, VA North Texas Healthcare System, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VISN 17, 10N17
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Bypass; Arteriosclerosis
Keywords: Coronary artery bypass; Stents; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Restenosis; Paclitaxel
MeSH Terms: conditions — Arteriosclerosis; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Express 2 bare metal stent
  Interventions: Device: Express 2 bare metal stent
- 2 (Experimental): Taxus, paclitaxel-eluting stent
  Interventions: Device: Taxus polymer-based paclitaxel-eluting stent

INTERVENTIONS:
Device: Taxus polymer-based paclitaxel-eluting stent — Two different types of stents (paclitaxel-eluting and a similar bare metal stent) are being compared in saphenous vein graft lesions.
  Other Names: Taxus drug-eluting stents
  Arms: 2
Device: Express 2 bare metal stent — Two different types of stents (paclitaxel-eluting and a similar bare metal stent) are being compared in saphenous vein graft lesions.
  Arms: 1

SUMMARY:
The main purpose of this study is to determine whether implantation of a paclitaxel-eluting stent (Taxus™) in saphenous vein graft lesions will reduce the incidence of in-stent restenosis after 12 months when compared to a similar bare metal stent.

DETAILED DESCRIPTION:
Introduction: The prevalence of coronary artery bypass graft (CABG) surgery is high in the veteran population. Saphenous veins are used as conduits in the majority of CABG operations. Compared to arterial conduits, saphenous vein grafts (SVGs) have a high rate of failure, requiring percutaneous coronary intervention (PCI) or repeat CABG. Bare metal stents are currently used in the majority of PCI in SVGs because they increase the procedural success rate and decrease restenosis. However, even with the use of bare metal stents, restenosis still occurs in 37-53% of the SVGs, often requiring repeat target vein graft revascularization.

Drug-eluting stents (DES) have been a major breakthrough in percutaneous coronary intervention because they significantly reduce the incidence of in-stent restenosis in de novo lesions of native coronary arteries. Even though, no randomized controlled trials have compared DES with bare stents in SVG interventions, DES are increasingly being used off label in this setting, based on registry data. DES are expensive and may not provide benefit in SVGs since the atherosclerotic process is different in SVGs and in native coronary arteries. We propose to compare the 12-month angiographic restenosis rates after implantation of a polymer-based paclitaxel-eluting stent or the Express-2 bare metal stent (which is identical to the paclitaxel-eluting stent but has no drug coating) in saphenous vein graft lesions.

Hypothesis: Compared to implantation of a bare metal stent, implantation of a similar paclitaxel-eluting stent (Taxus™, Boston Scientific, Nattick, Massachusetts) in saphenous vein graft lesion will reduce the incidence of angiographic in-stent restenosis after 12 months.

Specific objectives: We propose to randomize patients undergoing stenting of a saphenous vein graft lesion to a bare metal stent or an identical paclitaxel-eluting stent (Taxus™) in order to determine:

1. whether the paclitaxel-eluting stent will reduce the incidence of binary angiographic in-stent restenosis, as assessed by 12-month follow-up quantitative coronary angiography (primary study endpoint), and
2. whether the paclitaxel-eluting stent will reduce the 24-month incidence of ischemia-driven target vessel revascularization, target vessel failure, overall major adverse cardiac and cerebrovascular events, and intra-stent intimal hyperplasia accumulation, as measured by intravascular ultrasound (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* at least one 50-99% de-novo or restenotic lesion in a saphenous vein graft that is between 2.5 and 4.0 mm in diameter, requiring percutaneous coronary intervention according to the opinion of the attending cardiologist
* willing to return for repeat coronary angiography after 12 months
* able to give informed consent

Exclusion Criteria:

* previous or planned use of intravascular brachytherapy in the target vessel
* a left ventricular ejection fraction of less than 25 percent
* hemorrhagic diatheses
* contraindications or allergy to aspirin, thienopyridines, paclitaxel, or stainless steel
* a history of anaphylaxis in response to iodinated contrast medium
* use of paclitaxel within 12 months before study entry or current use of colchicine
* a serum creatinine level of more than 2.0 mg per deciliter (177 µmol per liter)
* a leukocyte count of less than 3500 per cubic millimeter, or a platelet count of less than 100,000 per cubic millimeter
* a recent positive pregnancy test, breast-feeding, or the possibility of a future pregnancy
* coexisting conditions that limit life expectancy to less than 24 months or that could affect a patient's compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
binary angiographic in-stent restenosis, as assessed by 12-month follow-up quantitative coronary angiography | 12 months

SECONDARY OUTCOMES:
intrastent intimal hyperplasia accumulation as measured by IVUS | 12 months for IVUS and 24 months for clinical follow-up
incidence of ischemia-driven target vessel revascularization, target vessel failure, and overall major adverse cardiac and cerebrovascular events at 24-month follow-up | 12 months for IVUS and 24 months for clinical follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — VA North Texas Health Care System, University of Texas Southwestern Medical School
Locations (5):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - VA Iowa City Healthcare system, Iowa City, Iowa
  - VA North Texas Health Care System, Dallas, Texas
  - Michael E. Debakey VA Medical Center, Houston, Texas
- Onassis Cardiac Surgery Center, Athens, Greece

REFERENCES:
- [Result] Brilakis ES, Lichtenwalter C, de Lemos JA, Roesle M, Obel O, Haagen D, Saeed B, Gadiparthi C, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger P, Banerjee S. A randomized controlled trial of a paclitaxel-eluting stent versus a similar bare-metal stent in saphenous vein graft lesions the SOS (Stenting of Saphenous Vein Grafts) trial. J Am Coll Cardiol. 2009 Mar 17;53(11):919-28. doi: 10.1016/j.jacc.2008.11.029. PMID 19281920
- [Result] Lichtenwalter C, de Lemos JA, Roesle M, Obel O, Holper EM, Haagen D, Saeed B, Iturbe JM, Shunk K, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger P, Banerjee S, Brilakis ES. Clinical presentation and angiographic characteristics of saphenous vein graft failure after stenting: insights from the SOS (stenting of saphenous vein grafts) trial. JACC Cardiovasc Interv. 2009 Sep;2(9):855-60. doi: 10.1016/j.jcin.2009.06.014. PMID 19778774
- [Result] Michael TT, Abdel-karim AR, Papayannis A, Lichtenwalter C, de Lemos JA, Obel O, Addo T, Roesle M, Haagen D, Rangan BV, Saeed B, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger PB, Banerjee S, Brilakis ES. Recurrent cardiovascular events with paclitaxel-eluting versus bare-metal stents in saphenous vein graft lesions: insights from the SOS (Stenting of Saphenous Vein Grafts) trial. J Invasive Cardiol. 2011 Jun;23(6):216-9. PMID 21646644
- [Result] Brilakis ES, Lichtenwalter C, Abdel-karim AR, de Lemos JA, Obel O, Addo T, Roesle M, Haagen D, Rangan BV, Saeed B, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger P, Banerjee S. Continued benefit from paclitaxel-eluting compared with bare-metal stent implantation in saphenous vein graft lesions during long-term follow-up of the SOS (Stenting of Saphenous Vein Grafts) trial. JACC Cardiovasc Interv. 2011 Feb;4(2):176-82. doi: 10.1016/j.jcin.2010.10.003. PMID 21349456
- [Result] Michael TT, Badhey N, Banerjee S, Brilakis ES. Comparison of characteristics and outcomes of patients undergoing saphenous vein graft stenting who were or were not enrolled in the stenting of saphenous vein grafts randomized controlled trial. J Investig Med. 2011 Feb;59(2):259-66. doi: 10.231/JIM.0b013e318207066c. PMID 21200334
- [Result] Badhey N, Lichtenwalter C, de Lemos JA, Roesle M, Obel O, Addo TA, Haagen D, Abdel-Karim AR, Saeed B, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger PB, Banerjee S, Brilakis ES. Contemporary use of embolic protection devices in saphenous vein graft interventions: Insights from the stenting of saphenous vein grafts trial. Catheter Cardiovasc Interv. 2010 Aug 1;76(2):263-9. doi: 10.1002/ccd.22438. PMID 20665875
- See also: Trial main website — http://www.northtexas.va.gov/research/SOS/index.asp